CLINICAL TRIAL: NCT05764954
Title: A Prospective Clinical Trial of Tumor Immunomodulation Using Tumor-Treating Fields (TTFields) in Patients With Early-Stage Resectable Lung Adenocarcinoma
Brief Title: A Study of Tumor-Treating Fields (TTFields) in People With Lung Adenocarcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-387
Record Dates: First submitted 2023-02-22; First posted 2023-03-13 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Adenocarcinoma of Lung
Keywords: NOVOTTF-200T system; TTFields treatment; 22-387
MeSH Terms: conditions — Adenocarcinoma of Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- NovoTTF-200T System Tumor-Treating Fields (TTFields) (Experimental): Following pathological confirmation on of lung ADC, patients will proceed with TTFields treatment. The NovoTTF-200T System is an investigational medical device delivering 150 kHz TTFields to the patient's chest. The device is applied continuously for an average duration of 18 hours per day for 3 weeks (+/- 1 week).
  Interventions: Device: NovoTTF-200T System

INTERVENTIONS:
Device: NovoTTF-200T System — The device is applied continuously for an average duration of 18 hours per day for 3 weeks (+/- 1 week).

SUMMARY:
The researchers are doing this study to find out if treatment with TTFields using the NovoTTF-200T System is safe and practical (feasible) before surgical removal (resection) of lung adenocarcinoma (ADC). The researchers will also look at how the treatment may help the body's immune system to fight cancer.

ELIGIBILITY:
Inclusion Criteria:

* The participant (or legally acceptable representative [LAR], if applicable) provides written informed consent for the study.
* The participant is ≥22 years of age on the day of signing informed consent.
* The participant has clinical stage 1A2, 1A3 or IB biopsy-proven lung ADC and is eligible for anatomical resection.
* The participant has a lung nodule >1 cm and suspected lung ADC with a plan to undergo biopsy.
* The participant with multiple nodules has one nodule that meets the criteria.
* The participant has no history of prior malignancy in the chest or has undergone potentially curative therapy with no evidence of that disease recurrence for 5 years since initiation of that therapy.

Exclusion Criteria:

* Patients receiving therapy for concurrent active malignancy
* Patients with a history of cardiac arrhythmias and/or pacemaker use
* Patients with lung nodules <1cm
* Patients with lung nodules that are pure ground glass opacities (GGOs) of any size
* Patients with lung nodules that are <50% solid of any size

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-08-04 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Adverse events, severity and frequency | 1 year
  based on Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Prasad Adusumilli, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Consent Only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent Only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent Only), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Consent Only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent Only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Consent Only), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm